CLINICAL TRIAL: NCT06877442
Title: Correlation of Neuronal Cytoskeletal Integrity With Severity of Symptoms and Cognitive Decline In Mood Disorders
Brief Title: Neurofilament Light Chain Correlation With Severity of Symptoms and Cognitive Decline in Mood Disorders
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, waleed ashraf hamdy ahmed, Doctor, Assiut University
Other Study IDs: NFL mood disorders
Record Dates: First submitted 2025-03-10; First posted 2025-03-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Mood Disorders
Keywords: mood disorders; neurofilament light chain
MeSH Terms: conditions — Mood Disorders; Charcot-Marie-Tooth disease, Type 1F

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- group A Patients with major depression: meet the Diagnostic And Statistical Manual Of Mental Disorders Fifth Edition (DSM-5) criteria for major depressive disorder they will undergo the following
  1. Hamilton depression rating scale
  2. montreal cognitive assessment c, serum level of neurofilament light chain
  Interventions: Diagnostic Test: serum level of neurofilament light chain
- group B Bipolar Disorder: meet the Diagnostic And Statistical Manual Of Mental Disorders Fifth Edition (DSM-5) criteria for Bipolar Disorder they will undergo the following
  1. young mania rating scale
  2. montreal cognitive assessment
  3. serum level of neurofilament light chain
  Interventions: Diagnostic Test: serum level of neurofilament light chain
- group C healthy control: not known to have any medical or mental illness they will undergo the following
  1. montreal cognitive assessment
  2. serum level of neurofilament light chain
  Interventions: Diagnostic Test: serum level of neurofilament light chain

INTERVENTIONS:
Diagnostic Test: serum level of neurofilament light chain — labarotory investigation to evaluate serum level of neurofilament light chain

SUMMARY:
* Explore correlation of neurofilament light chain serum level and severity of symptoms and cognitive impairment in mood disorders
* Explore How novel brain markers as neurofilament light chain can be useful in detection and prognosis of mood disorders

DETAILED DESCRIPTION:
Cytoskeletal integrity, represented by neurofilament light chain (NfL), has emerged as a critical biomarker for neuroaxonal injury, with growing evidence linking it to mood disorders such as major depressive disorder (MDD) and bipolar disorder (BD). Neurofilaments are structural proteins essential for maintaining neuronal stability, and NfL, the smallest subunit, is released into extracellular fluids like cerebrospinal fluid (CSF) and blood following neuronal damage. Recent advancements in immunoassay technologies have enabled the reliable quantification of NfL in peripheral blood, providing a minimally invasive method to assess brain pathology (1).

Mood disorders are characterized by structural brain alterations, including reduced white matter integrity and gray matter volume loss, suggesting underlying neuroaxonal damage. Elevated blood NfL levels have been reported in patients with Major Depressive Disorder and Bipolar Disorder , with increases ranging from 1.2 to 2.5-fold compared to healthy controls, indicating a potential link between cytoskeletal disruption and mood disorder pathology (1,2).

In MDD, higher NfL levels have been associated with cognitive dysfunction and white matter abnormalities, highlighting the role of cytoskeletal integrity in disease severity (3).

Similarly, in Bipolar Disorder, elevated NfL levels have been linked to cognitive deficits and structural brain changes, particularly during acute episodes, further supporting the involvement of neuroaxonal injury in mood disorder progression (2,4).

However, the interpretation of NfL levels in mood disorders is complicated by factors such as age, body mass index (BMI), and cardiovascular risk factors, which influence NfL variability (1). Despite these challenges, NfL holds promise as a biomarker for assessing cytoskeletal integrity and monitoring disease progression in mood disorders, offering new insights into their neurobiological underpinnings. Further research is needed to elucidate the mechanisms driving NfL release and its clinical utility in psychiatric practice.

ELIGIBILITY:
Participants will be divided into three groups (A) Patients with Major depressive episode (B) Patients with Bipolar Disorder Manic Episode

1. Inclusion criteria:

   1. age 15-50 years old
   2. both sexes will be included
   3. meet the Diagnostic And Statistical Manual Of Mental Disorders Fifth Edition (DSM-5) criteria for major depressive disorder or Bipolar disorder
2. Exclusion criteria:

   1. Major Medical or Neurological Diseases.
   2. History of Traumatic Brain Injury, Major Fracture.
   3. Alcohol or Substance Use Disorder. (C) Healthy control

a. Inclusion criteria:

1. age- and sex-matching with group A, B
2. Healthy Control without any of major physical conditions or psychiatric disorder

Ages: 15 Years to 50 Years | Sex: All
Age Groups: Child, Adult
Study Population: Participants will be divided into three groups (A) Patients with Major depressive episode (B) Patients with Bipolar Disorder Manic Episode (C) Healthy control thirty participants in each group from 15-50 years old amtching in age and sex with each group
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
correlation of neurofilament light chain with severity of symptoms in mood disorders | baseline
  correlation of serum level of neurofilament light chain and severity of symptoms in mood disorders
correlation of neurofilament light chain with cognitive function in mood disorders | baseline
  correlation of serum level of neurofilament light chain and cognitive functions in mood disorders

CONTACTS AND LOCATIONS:
Overall Officials: Wageeh A Hassan, Study Chair — Assiut University; Hossam E Khalifa, Study Director — Assiut University

REFERENCES:
- [Background] Bavato F, Barro C, Schnider LK, Simren J, Zetterberg H, Seifritz E, Quednow BB. Introducing neurofilament light chain measure in psychiatry: current evidence, opportunities, and pitfalls. Mol Psychiatry. 2024 Aug;29(8):2543-2559. doi: 10.1038/s41380-024-02524-6. Epub 2024 Mar 19. PMID 38503931
- [Background] Jakobsson J, Bjerke M, Ekman CJ, Sellgren C, Johansson AG, Zetterberg H, Blennow K, Landen M. Elevated concentrations of neurofilament light chain in the cerebrospinal fluid of bipolar disorder patients. Neuropsychopharmacology. 2014 Sep;39(10):2349-56. doi: 10.1038/npp.2014.81. Epub 2014 Apr 3. PMID 24694925
- [Background] Bavato F, Cathomas F, Klaus F, Gutter K, Barro C, Maceski A, Seifritz E, Kuhle J, Kaiser S, Quednow BB. Altered neuroaxonal integrity in schizophrenia and major depressive disorder assessed with neurofilament light chain in serum. J Psychiatr Res. 2021 Aug;140:141-148. doi: 10.1016/j.jpsychires.2021.05.072. Epub 2021 Jun 2. PMID 34116440
- [Background] Aggio V, Fabbella L, Finardi A, Mazza EB, Colombo C, Falini A, Benedetti F, Furlan R. Neurofilaments light: Possible biomarker of brain modifications in bipolar disorder. J Affect Disord. 2022 Mar 1;300:243-248. doi: 10.1016/j.jad.2021.12.122. Epub 2021 Dec 31. PMID 34979181